CLINICAL TRIAL: NCT05465980
Title: Development and Validation of the Prediction Model for Cognitive Impairment in Elderly Patients After Acute Ischemic Stroke
Brief Title: Development and Validation of the Prediction Model for Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20223357018
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the "Chinese Stroke Report" released in 2020, the incidence of stroke in China is 1114.8/100,000, acute ischemic stroke (AIS) accounts for 70% to 80% of the total number of stroke population, and elderly stroke patients are up to 2/3. About 1/3 of stroke patients would experience post-stroke cognitive impairment (PSCI), which seriously affected patients' quality of life and survival time, and increases disease and economic burden. Therefore, early identification, assessment, prevention and intervention of PSCI, and improvement of patients' quality of life and prognosis have become the focus of clinical research.

This is a prospective cohort study. We intend to: (1) continuously collect elderly AIS patients who will be admitted to the Department of Neurology, The Department of Rehabilitation and the Department of Gerontology of Shenzhen Second People's Hospital from 2022 year to 2024 year; (2) collect baseline and follow-up data, and build a prediction model for cognitive impairment in elderly AIS patients; (3) internal validation using Bootstrap model; (4) collect the data of the elderly AIS patients who will be admitted to Shenzhen Longhua District People's Hospital andShenzhen Longgang Central Hospital, and conduct external validation; (5) evaluate the predictive efficacy of the model.

DETAILED DESCRIPTION:
This study consists of two parts. The first part is to develop a predictive model for cognitive impairment in elderly patients with acute ischemic stroke. Continuously collect the baseline data and follow-up data of elderly AIS patients admitted to the Shenzhen Second People's Hospital from September 2022 to December 2023, including general demographic data, laboratory examination indicators, imaging indicators and assessment scales. Take the occurrence of PSCI as the dependent variable and the risk factors of PSCI in elderly AIS patients will be analyzed. Multivariate Cox regression will be used to develop a prediction model for cognitive impairment in elderly AIS patients.

The second part is to do clinical evaluation of prediction model of cognitive impairment in elderly patients with acute ischemic stroke. Bootstrap method will be used for internal validation of the model. Continuously collect the data of elderly AIS patients from January 2024 to December 2024 from the other two hospitals in Guangdong Province, China. Externally validate the model and evaluate the clinical application effect of PSCI prediction model in elderly AIS patients using C-index, reclassification index, calibration curve, time-dependent ROC curve and other indicators. Finally, the model is presented by nomogram.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 60 years or older.
2. Stroke occurring within 7 days.
3. Meet the diagnostic criteria of Chinese Guidelines for the Diagnosis and Treatment of Acute ischemic Stroke 2018.
4. Informed consent.

Exclusion Criteria:

1. Incomplete main clinical data;
2. Patients with transient ischemic attack;
3. Patients had cognitive dysfunction before enrollment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The elderly patients with acute ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 496 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
MMSE score | From July 1, 2022 to May 31, 2025
  The primary outcome will be assessed by the Mini-mental State Examination(MMSE) scale

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Xie, master, Principal Investigator — Shenzhen Second People's Hospital

IPD SHARING:
Plan to Share IPD: No